CLINICAL TRIAL: NCT01765101
Title: Therapeutic Effects of Ready-made Full-length Lateral Wedged Insoles and Customized Full-length Lateral Wedged Insoles on Patients With Knee Osteoarthritis : a Double Blind, Randomized Controlled Study
Brief Title: Therapeutic Effects of Insoles on Patients With Knee Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, MD, Associate professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SKH-8302-102-DR-32
Record Dates: First submitted 2013-01-04; First posted 2013-01-10 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; therapeutic effect; insole
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- customized insoles (Experimental): customized full-length lateral wedged shoe insoles
  1 month and 3 months study the immediate, short-term and intermediate-term therapeutic effects
  Interventions: Other: customized insoles
- ready made insoles (Placebo Comparator): ready-made full-length lateral wedged shoe insoles at 1 and 3 months
  study the immediate, short-term and intermediate-term therapeutic effects
  Interventions: Other: ready made insoles

INTERVENTIONS:
Other: customized insoles — To study the immediate, short-term and intermediate-term therapeutic effects, including psychological function, physical activity , functional performance and quality of life, physical functional ability, pain and balance performance
  Other Names: customized full-length lateral wedged insoles: ICB
  Arms: customized insoles
Other: ready made insoles — To study the immediate, short-term and intermediate-term therapeutic effects, including psychological function, physical activity , functional performance and quality of life, physical functional ability, pain and balance performance
  Other Names: ready made full-length lateral wedged insoles: La New
  Arms: ready made insoles

SUMMARY:
Using double blind, randomized controlled design to study the immediate, short-term and intermediate-term therapeutic effects of ready-made full-length lateral wedged shoe insoles and customized full-length lateral wedged shoe insoles to patients with knee osteoarthritis, under the basis of International Classification Functioning, Disability and Health.

DETAILED DESCRIPTION:
A total of 90 patients will be collected. The participants will be randomized into two groups, including ready-made full-length lateral wedged shoe insoles group and customized full-length lateral wedged shoe insoles group. The psychological function (Hospital anxiety and depression scale, Graded chronic pain scale, Multidimensional fatigue inventory, Fear-avoidance belief questionnaire), physical activity (CHAMPS physical activity questionnaire), functional performance (Western Ontario and McMaster Universities Osteoarthritis index、Knee injury and Osteoarthritis Outcome Score) and quality of life (World Health Organization-Quality of life-Brief Vision、Osteoarthritis Quality of Life、Osteoarthritis- Knee and Hip Quality of Life) will be evaluated. Physical functional ability (10 meter normal and fast walk, up and down stairs, and 5 repeated chair-rising time), pain (Visual analog scale, pain pressure threshold ) and balance performance (static postural stability and dynamic stability by Biodex Stability System, including postural stability, dynamic limits of stability and fall risk) will be evaluated before and immediately after the ready-made full-length shoe insoles and customized full-length shoe insoles are prescribed. All the evaluations, including physical functional ability, pain, balance, psychological, physical activity, functional performance, and quality of life, will be re-evaluated at one month after and three months after modified shoe insoles wearing. Subjects and evaluator were both blinded to the group's classification during the whole course of study.

ELIGIBILITY:
Inclusion Criteria:

* fulfill the combined clinical and radiographic criteria for knee osteoarthritis, as established by the American College of Rheumatology
* with Kellgren-Lawrence scores of 2 or higher in the isolated medial compartment

Exclusion Criteria:

* with a history of previous knee surgery with an implant
* reduced lateral compartment and/or combined medial and lateral compartments in knee joints were excluded
* pregnant or planning to become pregnant
* self-reported history of vertigo, malignancy, stroke, or other conditions that may impair vestibular function

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
pain | change from baseline at one month and three months after modified shoe insoles wearing
  Visual analog scale, pain pressure threshold

SECONDARY OUTCOMES:
Physical functional ability | change from baseline at one month and three months after modified shoe insoles wearing
  10 meter normal and fast walk, up and down stairs, and 5 repeated chair-rising time
psychological function | change from baseline at one month and three months after modified shoe insoles wearing
  Hospital anxiety and depression scale, Graded chronic pain scale, Multidimensional fatigue inventory, Fear-avoidance belief questionnaire
functional performance | change from baseline at one month and three months after modified shoe insoles wearing
  Western Ontario and McMaster Universities Osteoarthritis index、Knee injury and Osteoarthritis Outcome Score
quality of life | change from baseline at one month and three months after modified shoe insoles wearing
  World Health Organization-Quality of life-Brief Vision、Osteoarthritis Quality of Life、Osteoarthritis- Knee and Hip Quality of Life
balance performance | change from baseline at one month and three months after modified shoe insoles wearing
  static postural stability and dynamic stability by Biodex Stability System, including postural stability, dynamic limits of stability and fall risk
physical activity | change from baseline at one month and three months after modified shoe insoles wearing
  CHAMPS physical activity questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital; Taipei Medical University
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan, Taiwan